CLINICAL TRIAL: NCT05948020
Title: Efficacy and Safety of Orally Administered Engineered Probiotics (CBT102-A) for the Treatment of Children With Phenylketonuria：a Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study
Brief Title: Efficacy and Safety of Orally Administered Engineered Probiotics (CBT102-A) for the Treatment of Children With Phenylketonuria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Hedu Biotechnology (Shanghai) Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT-102
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-07

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking to the investigation sites and subjects (including subjects' guardians)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT102-A group (Experimental): 10 subjects receive oral CBT102-A with three meals per day for a total of 20 days
  Interventions: Biological: CBT102-A capsule
- Placebo group (Placebo Comparator): 5 subjects receive oral placebo with three meals per day for a total of 20 days
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Biological: CBT102-A capsule — Orally CBT102-A will be supplied by CommBio Therapeutics. It is an enteric-coated capsule with 1.25×10^11 live cell. The shelf life is 6 months.
  Subjects receive oral dose of 1 capsule CBT102-A (1.25 x 10^11 live cell) before three meals per day on Day 1 to Day 4; Subjects receive oral dose of 2 capsule CBT102-A (2.5 x 10^11 live cell) before three meals per day on Day 5 to Day 8; Subjects receive oral dose of 4 capsule CBT102-A (5 x 10^11 live cell) before three meals per day on Day 9 to Day 12; Subjects receive oral dose of 8 capsule CBT102-A (1 x 10^12 live cell) before three meals per day on Day 13 to Day 20; All subjects will be observed for 3 days (Day 21~Day 23) without intervene in hospital and will be followed up weekly for 4 consecutive weeks after discharge（Day 51）.
  Arms: CBT102-A group
Other: Placebo capsule — Orally placebo will be supplied by CommBio Therapeutics. It is an enteric-coated capsule with Lactose powder filler. The shelf life is 6 months. The color, condition, smell and other appearances are exactly the same as CBT102-A.
  Subjects receive oral dose of 1 capsule placebo before three meals per day on Day 1 to Day 4; Subjects receive oral dose of 2 capsule placebo before three meals per day on Day 5 to Day 8; Subjects receive oral dose of 4 capsule placebo before three meals per day on Day 9 to Day 12; Subjects receive oral dose of 8 capsule placebo before three meals per day on Day 13 to Day 20; All subjects will be observed for 3 days (Day 21~Day 23) without intervene in hospital and will be followed up weekly for 4 consecutive weeks after discharge（Day 51）.
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study. A total of 15 children with phenylketonuria(PKU) age 3 to 17 years will be randomized to two groups. Experimental group of 10 children will intervene engineered probiotics (CBT102-A) for 20 days and 5 children will intervene placebo. The goal of this study is to determine whether CBT102-A is an effective and safe treatment for PKU.

DETAILED DESCRIPTION:
Due to an increased blood phenylalanine (Phe) concentration, untreated children with PKU will develop progressively intellectual disability. Engineered probiotics can metabolize Phe into other products in the intestine by expressing related exogenous proteins in the Phe metabolic pathway, thereby reducing Phe concentration in the intestine and blood.

Animal experiments have confirmed the efficacy and safety of CBT102-A. This study will enroll children with PKU age 3 to 17 years according to a strict inclusion and exclusion criteria. Subjects who meet the requirements will be randomly assigned on Day 1 and start the study administration. The administration period of both groups is 20 days (Day 1~Day 20), in which the experimental group receives CBT102-A with 4 dose levels, and the control group receives placebo administration, with the same mode, frequency, time, cycle and dose as the experimental group. All subjects will be observed for 3 days (Day 21~Day 23) without intervene in hospital and will be followed up weekly for 4 consecutive weeks after discharge（Day 51）.

Change of blood Phe concentration and occurrence of Treatment-Emergent Adverse Events(TEAE) with PKU will be used to evaluate the efficacy and safety of the CBT102-A.

ELIGIBILITY:
Inclusion Criteria:

* Blood phe ≥ 600μmol/L at newborn screening;
* Blood phe ≥ 600μmol/L at least 3 times in the last 1 year before screening, and the blood Phe ≥ 600μmol/L in the last 1 time;
* Screening laboratory evaluations (e.g., chemistry panel, complete blood count, urinalysis, creatinine clearance, CRP) within normal limits or judged to be not clinically significant by the investigator;
* Stable diet for at least 60 days prior to screening;
* Able to produce at least 2 bowel movements per week on average without using any form of laxatives;
* Adolescents and children's guardians can voluntarily complete the whole process of informed consent, including stool, urine and blood collection, adherence to diet control, hospital monitoring, follow-up and oral trial drug compliance, and sign informed consent.

Exclusion Criteria:

* The standard percentile values of height and weight of Chinese children aged 0 to 18 years were evaluated with weight less than P3 or weight greater than P97；
* History of active or chronic passage of 3 or more loose stools per day；
* Have any medical conditions or medications that may affect the absorption of medications or nutrients；
* History of or current immunodeficiency disorder including autoimmune disorders；
* Subjects with obvious influenza-like symptoms caused by COVID-19 or other viral infections during screening；
* Hepatitis B surface antigen and/or hepatitis C antibodies and/or treponema pallidum antibodies positive；
* Subjects who are dependent on drugs and alcohol；
* Received gene therapy related to PKU；
* Intolerant or allergic to Escherichia coli Nissle 1917 (EcN)；
* Active gastrointestinal bleeding or a proven history of gastrointestinal bleeding within 60 days prior to screening；
* Antibiotics within 28 days before the planned first dose of investigational product (IP), or anticipated during the study period；
* Take probiotic supplements within 28 days before the planned first dose of IP, or anticipated during the study period；
* A history of fever, confirmed bacteremia, or other active infection within 30 days prior to the planned first dose of IP；
* Drugs that use of the digestive system has been used within 30 days prior to the planned first dose of IP;
* Drugs that may affect gastrointestinal function has been used within 30 days prior to the planned first dose of IP;
* Major survery performed within 90 days before the anticipated first dose of IP or planned surgery or hospitalization during the study period；
* Take sapropterin (KUVAN®) within 1 week before the planned first dose of IP；
* Use pegylated recombinant phenylalanine ammonia lyase (PALYNZIQ™) within 30 days before the planned first dose of IP；
* History of severe immune adverse reactions to PALYZIQ；
* Participated in an interventional clinical trial and used the investigational drug within 60 days or 5 half-lives before the planned first dose of IP；
* Subjects who may not be able to complete the study for other reasons.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-09-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Blood Phe Concentration | From baseline to Day 51
  This is a repeatedly measures outcome; Blood Phe concentration will be detected at baseline, administration(Day 1~Day 20), observation(Day 21~Day 23) and follow-up periods(Day 51); During the administraion time, Phe concentrations will be measured at 4 hours after each day on Day 4,Day 8, Day 12, Day 15, Day 18, Day 20; A drop of blood will be collected from the end of the finger on the filter paper and will be detected by tandem mass spectrometry.

SECONDARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events（TEAE）≥2 Grade | From baseline to Day 23
  The grade of TEAE will be assessed according to Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0; TEAE ≥ 2 grade define as occurrence of age-appropriate limitations in instrumental activities of daily living; Adverse events require medical intervention.
Occurrence of TEAE | From baseline to Day 51
  All treatment emerged adverse events during the whole study
Changing Value of Subjects Urinary Metabolites | From baseline to Day 23
  This is a repeatedly measures outcome; During the administraion time, subjects' urine will be collected after each day on Day 8, Day 12, Day 20 and Day 23; The changes of metabolites will be detected by tandem mass spectrometry.
Changing Value of Subjects Fecal Metabolites | From baseline to Day 23
  This is a repeatedly measures outcome; During the administraion time, subjects' fecal will be collected after each day on Day 8, Day 12, Day 20 and Day 23; The changes of metabolites will be detected by tandem mass spectrometry.
Clearance of CBT102-A from Fecal | From baseline to Day 23
  This is a repeatedly measures outcome; CBT102-A transit through the gastrointestinal tract will be measured with fecal quantitative polymerase chain reaction (qPCR) assays from fecal samples collected at baseline,Day 20 and Day 23 during the dosing period; CBT102-A clearance reflects a test value of below the limit of quantitation (BLQ) occurring after the indicated number of days following the last dose of investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Principal Investigator — Children's Hospital of Fudan University; Huijun Wang, Principal Investigator — Children's Hospital of Fudan University; Haitao Zhu, Principal Investigator — Children's Hospital of Fudan University; Yajie Su, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No